CLINICAL TRIAL: NCT00633893
Title: A Safety and Efficacy Trial Evaluating the Use of Apixaban for the Extended Treatment of Deep Vein Thrombosis and Pulmonary Embolism
Brief Title: Efficacy and Safety Study of Apixaban for Extended Treatment of Deep Vein Thrombosis or Pulmonary Embolism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV185-057; EUDRACT: 2007-004953-27
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 2.5 mg
  Interventions: Drug: Apixaban
- 2 (Experimental): 5.0 mg
  Interventions: Drug: Apixaban
- 3 (Active Comparator): 0 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban — Tablets, Oral, twice daily, 12 months
  Other Names: BMS-562247
  Arms: 1; 2
Drug: Placebo — Tablets, Oral, twice daily, 12 months
  Arms: 3

SUMMARY:
The purpose is to evaluate the effects of an investigational blood thinner, apixaban, in preventing venous thromboembolic (VTE) recurrence or death in patients who have completed their intended treatment for deep vein thrombosis (DVT) or pulmonary embolism (PE)

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age;
* Clinical diagnosis of Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE);
* Anticoagulant treatment completed
* No recurrence of Venous Thromboembolism (VTE)

Exclusion Criteria:

* Subjects with indications for long-term treatment with a vitamin K antagonist
* Active bleeding or high risk for serious bleeding
* Short life expectancy
* Uncontrolled high blood pressure
* Impaired kidney or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2711 (Actual)
Dates: Start 2008-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (349):
- United States (87):
  - Alabama Clinical Therapeutics, Llc, Birmingham, Alabama
  - Cardiovascular Consultants, Ltd., Phoenix, Arizona
  - Robert J. Bloomberg, Md, Pc, Tempe, Arizona
  - Fort Smith Lung Center, Fort Smith, Arkansas
  - Beaver Medical Group, Banning, California
  - Scripps Clinic/Scripps Health And Green Hospital, La Jolla, California
  - Healthcare Partners Medical Group, Los Angeles, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Desert Med Grp Inc, Dba Desert Oasis Healthcare Med Group, Palm Springs, California
  - Indus Clinical Research Institute, Inc., Pomona, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Harbor Ucla Medical Center, Torrance, California
  - Progressive Clinical Research, Vista, California
  - Rocky Mountain Internal Medicine, Aurora, Colorado
  - New West Physicians, Golden, Colorado
  - Alfieri Cardiology, Newark, Delaware
  - Bay Pines Va Healthcare Systems, Bay Pines, Florida
  - Research Alliance, Inc., Clearwater, Florida
  - St. Francis Sleep Allergy & Lung Institute, Clearwater, Florida
  - Berma Research Group, Fort Lauderdale, Florida
  - Healthworx, Hollywood, Florida
  - Hematology Oncology Associates, Loxahatchee Groves, Florida
  - South Miami Heart Center, Miami, Florida
  - Physicians Regional Medical Group, Naples, Florida
  - Richard A. Mclean M.D., P.A., Plantation, Florida
  - Tampa Clinical Research, Tampa, Florida
  - Primary Care Of The Treasure Coast, Inc., Vero Beach, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Vascular Surgical Associates, Pc, Austell, Georgia
  - Atlanta Institute For Medical Research, Inc, Decatur, Georgia
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - Boise Orthopedic Clinic, Boise, Idaho
  - Saltzer Medical Group, Nampa, Idaho
  - Infectious Disease Of Indiana Psc, Carmel, Indiana
  - Office Of:Eugene C. Fletcher, Md, New Albany, Indiana
  - Heartland Vascular Medicine And Surgery, Windsor Heights, Iowa
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Owensboro Heart & Vascular, Owensboro, Kentucky
  - Pen Bay Medical Center, Rockport, Maine
  - Anne Arundel Health System Research Institute, Inc., Annapolis, Maryland
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Veterans Affairs Medical Center, Kansas City, Missouri
  - Mercury Street Medical Group, Pllc, Butte, Montana
  - Great Falls Clinic, Llp, Great Falls, Montana
  - Internal Medical Associates Of Grand Island, P.C, Grand Island, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Kaleida Health System, Buffalo, New York
  - Goshen Medical Associates, Goshen, New York
  - Sjh Cardiology Associates, Liverpool, New York
  - Richmond University Medical Center, Staten Island, New York
  - New York Medical College, Valhalla, New York
  - Thomas L. Ortel, Md, Phd, Durham, North Carolina
  - Valley Internal Medicine, Fayetteville, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Whiteville Medical Associates, P.A., Whiteville, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Remington Davis Inc., Columbus, Ohio
  - Jobst Vascular Center At The Toledo Hospital, Toledo, Ohio
  - Cor Clinical Research, Llc, Oklahoma City, Oklahoma
  - Pma Medical Specialists, Phoenixville, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Charleston Hematology Oncology Associates, Pa, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Three Rivers Medical Associates, Pa, Irmo, South Carolina
  - Clinical Research Authority, Llc, Murrells Inlet, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Amarillo Heart Clinical Research Institute Inc., Amarillo, Texas
  - Corsicana Medical Research, Corsicana, Texas
  - Ankur Doshi, Md, Houston, Texas
  - Northwest Heart Center, Tomball, Texas
  - Tanner Clinic, Layton, Utah
  - University Of Utah Hospital, Salt Lake City, Utah
  - University Of Virginia Health System, Charlottesville, Virginia
  - Sentara York Clinical Research, Norfolk, Virginia
  - Lake Washington Vascular, Pllc, Bellevue, Washington
  - Franciscan Research Center, Tacoma, Washington
  - Medical Assoicates Inc., Menomonee Falls, Wisconsin
- Argentina (11):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, Corrientes, Corrientes Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
- Australia (18):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Launceston, Tasmania
  - Local Institution, Box Hill, Victoria
  - Local Institution, Clayton, Victoria
  - Local Institution, Footscray, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Richmond, Victoria
  - Local Institution, Ringwood East, Victoria
  - Local Institution, Windsor, Victoria
  - Local Institution, Perth, Western Australia
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Vienna
- Brazil (13):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Brasília, Federal District
  - Local Institution, Belo Horizonte - Mg, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Rio Janeiro, Rio de Janeiro
  - Local Institution, Port Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Campinas, São Paulo
  - Local Institution, Santo Andre - Sp, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (11):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Pointe-Claire, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saint-Jérôme, Quebec
- Chile (5):
  - Local Institution, Punta Arenas, Magallanes Antartica
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Independencia, Santiago Metropolitan
  - Local Institution, Santiago, Santiago Metropolitan
- Czechia (7):
  - Local Institution, Kladno
  - Local Institution, Litomyšl
  - Local Institution, Městec Králové
  - Local Institution, Ostrava Vitkovice
  - Local Institution, Pilsen
  - Local Institution, Prague
  - Local Institution, Ústí nad Orlicí
- Denmark (9):
  - Local Institution, Arhus C
  - Local Institution, Brædstrup
  - Local Institution, Esbjerg
  - Local Institution, Frederiksberg
  - Local Institution, Hellerup
  - Local Institution, Herning
  - Local Institution, Hilleroed
  - Local Institution, Næstved
  - Local Institution, Silkeborg
- France (15):
  - Local Institution, Arras
  - Local Institution, Besançon
  - Local Institution, Brest
  - Local Institution, Clamart
  - Local Institution, Clermont-Ferrand
  - Local Institution, Dijon
  - Local Institution, Grenoble
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Saint-Priest-en-Jarez
  - Local Institution, Toulouse
  - Local Institution, Vernon
- Germany (15):
  - Local Institution, Berlin
  - Local Institution, Bochum
  - Local Institution, Bonn
  - Local Institution, Cologne
  - Local Institution, Dortmund
  - Local Institution, Dresden
  - Local Institution, Erfurt
  - Local Institution, Frankfurt
  - Local Institution, Göttingen
  - Local Institution, Karlsbad
  - Local Institution, Krefeld
  - Local Institution, Ludwigshafen
  - Local Institution, Mannheim
  - Local Institution, Munich
  - Local Institution, München
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, Shatin, N.T
- India (14):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Gurgaon, Haryana
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Bengaluru, Karnataka
  - Local Institution, Kochi, Kerala
  - Local Institution, Pune, Maharashtra
  - Local Institution, New Dehli, New Dehli
  - Local Institution, Mohali, Punjab
  - Local Institution, Ludhiana, Tagore Nagar
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Ahmedabad
  - Local Institution, Bangalore
  - Local Institution, Chennai
- Israel (13):
  - Local Institution, Afula
  - Local Institution, Giv‘atayim
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Kiryat Hadassah
  - Local Institution, Nahariya
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
- Italy (21):
  - Local Institution, Bollate
  - Local Institution, Bologna
  - Local Institution, Chieti Scalo
  - Local Institution, Cosenza
  - Local Institution, Ferrara
  - Local Institution, Florence
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Palermo
  - Local Institution, Pavia
  - Local Institution, Perugia
  - Local Institution, Piacenza
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Rozzano (Mi)
  - Local Institution, San Daniele Del Friuli (Ud)
  - Local Institution, Udine
  - Local Institution, Venezia
  - Local Institution, Vicenza
  - Local Institution, Vittorio Veneto (Tv)
- Mexico (14):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Puebla City, Puebla
  - Local Institution, Querétaro City, Querétaro
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Xalapa, Veracruz
- Norway (6):
  - Local Institution, Ålesund
  - Local Institution, Fredrikstad
  - Local Institution, Gjettum
  - Local Institution, Gjøvik
  - Local Institution, Hamar
  - Local Institution, Oslo
- Philippines (4):
  - Local Institution, Cavite
  - Local Institution, Davao City
  - Local Institution, Pasig
  - Local Institution, Quezon City
- Poland (13):
  - Local Institution, Arkonska 4
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Gdansk
  - Local Institution, Gdynia
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Przeworsk
  - Local Institution, Szczecin
  - Local Institution, Tarnobrzeg
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Portugal (2):
  - Local Institution, Guarda
  - Local Institution, Lisbon
- Local Institution, San Juan, Puerto Rico
- Romania (3):
  - Local Institution, Baia Mare
  - Local Institution, Bucharest
  - Local Institution, Târgu Mureş
- Russia (11):
  - Local Institution, Arkhangelsk
  - Local Institution, Kemerovo
  - Local Institution, Moscow
  - Local Institution, Novosibirsk
  - Local Institution, Rostov-on-Don
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Saratov
  - Local Institution, Tomsk
  - Local Institution, Yaroslavl
- Local Institution, Singapore, Singapore
- South Africa (10):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Centurion, Gauteng
  - Local Institution, Parktown, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Pietermaritzburg, KwaZulu-Natal
  - Local Institution, Bellville, Western Cape
  - Local Institution, George, Western Cape
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Worcester, Western Cape
- South Korea (3):
  - Local Institution, Busan
  - Local Institution, Jongno-Gu
  - Local Institution, Seoul
- Spain (17):
  - Local Institution, Torrevieja, Alicante
  - Local Institution, Badalona, Barcelona
  - Local Institution, Majadahonda, Madrid
  - Local Institution, San Sebastián de los Reyes, Madrid
  - Local Institution, Cadiz
  - Local Institution, Getafe
  - Local Institution, Girona
  - Local Institution, L'Hospitalet de Llobregat
  - Local Institution, León
  - Local Institution, Madrid
  - Local Institution, Mourente
  - Local Institution, Pamplona
  - Local Institution, Salamanca
  - Local Institution, Sant Boi de Llobregat
  - Local Institution, Tarragona
  - Local Institution, Toledo
  - Local Institution, Valencia
- Ukraine (11):
  - Local Institution, Chernihiv
  - Local Institution, Dnipropetrovsk
  - Local Institution, Donetsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
  - Local Institution, Lviv
  - Local Institution, Odesa
  - Local Institution, Ternopil
  - Local Institution, Vinnytsia
  - Local Institution, Zaporizhzhia
- United Kingdom (9):
  - Local Institution, Aberdeen, Aberdeenshire
  - Local Institution, Romford, Essex
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Hull, Humberside
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Bury St Edmunds, Suffolk
  - Local Institution, Coventry, West Midlands
  - Local Institution, Dudley, West Midlands

REFERENCES:
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Liu X, Thompson J, Phatak H, Mardekian J, Porcari A, Johnson M, Cohen AT. Extended anticoagulation with apixaban reduces hospitalisations in patients with venous thromboembolism. An analysis of the AMPLIFY-EXT trial. Thromb Haemost. 2016 Jan;115(1):161-8. doi: 10.1160/TH15-07-0606. Epub 2015 Oct 8. PMID 26446706
- [Derived] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant, first visit: 16 May 2008; Last participant, last visit: 24 August 2012.
Pre-assignment Details: 2711 enrolled/2482 randomized: 133 did not meet inclusion, exclusion criteria; 48 withdrew consent; 8 non-compliance; 3 each administrative and clinical reasons; 2 lost to follow up; 1 death; 1 adverse event (AE), 30 other. Data from 4 participants in site 0650 not analyzed/included in randomized population because source for data not confirmed.
Groups:
- Apixaban 2.5 mg: Participants received 2.5 mg oral tablet apixaban twice a day (BID)
- Apixaban 5 mg: Participants received 5 mg oral tablet apixaban BID.
- Placebo: Participants received matching placebo oral tablet BID.
Period: Overall Study
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Started | 840 | 813 (2 participants were randomized to 5 mg study drug but not treated.) | 829 (3 participants were randomized to placebo but not treated.)
Completed | 726 | 684 | 641
Not Completed | 114 | 129 | 188
Not completed — Death | 1 | 3 | 9
Not completed — Adverse Event | 65 | 58 | 126
Not completed — Withdrawal by Subject | 7 | 12 | 6
Not completed — Lost to Follow-up | 2 | 4 | 8
Not completed — Poor/non-compliance | 5 | 12 | 3
Not completed — Pregnancy | 2 | 1 | 1
Not completed — Not meet/no longer meets criteria | 4 | 6 | 4
Not completed — Other | 28 | 33 | 31

BASELINE CHARACTERISTICS:
Population: All randomized participants regardless of whether treatment was actually received were included; intent to treat (ITT) principle.
Groups:
- Apixaban 2.5 mg: Participants received 2.5 mg oral tablet apixaban BID.
- Total: Total of all reporting groups
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo | Total
Number analyzed (Participants) | 840 | 813 | 829 | 2482
Age Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.3) | 56.4 (15.6) | 57.1 (15.2) | 56.7 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 353 | 344 | 361 | 1058
  Male | 487 | 469 | 468 | 1424
Region of Enrollment [Number; unit: participants]
  Portugal | 1 | 1 | 0 | 2
  United States | 88 | 75 | 96 | 259
  Philippines | 5 | 3 | 3 | 11
  Hong Kong | 4 | 3 | 4 | 11
  Spain | 27 | 25 | 26 | 78
  Ukraine | 87 | 77 | 88 | 252
  Chile | 2 | 1 | 2 | 5
  Russian Federation | 45 | 49 | 46 | 140
  Israel | 34 | 34 | 34 | 102
  Italy | 67 | 65 | 61 | 193
  India | 24 | 23 | 24 | 71
  France | 60 | 55 | 50 | 165
  Australia | 30 | 28 | 31 | 89
  Denmark | 47 | 58 | 42 | 147
  South Africa | 34 | 42 | 30 | 106
  Korea, Republic of | 4 | 3 | 2 | 9
  Austria | 12 | 8 | 11 | 31
  United Kingdom | 33 | 29 | 30 | 92
  Czech Republic | 43 | 49 | 48 | 140
  Mexico | 22 | 18 | 22 | 62
  Canada | 22 | 17 | 15 | 54
  Argentina | 7 | 9 | 6 | 22
  Poland | 45 | 44 | 48 | 137
  Brazil | 19 | 24 | 30 | 73
  Singapore | 1 | 2 | 3 | 6
  Romania | 6 | 7 | 7 | 20
  Norway | 9 | 9 | 10 | 28
  Germany | 62 | 55 | 60 | 177
Index Event Classification [Number; unit: participants] — Number of participants with Proximal DVT (defined at the site) and number with PE (defined at the site). In the event a participant had both proximal DVT and PE, the participant was classified to PE.
  participants
    Proximal DVT | 544 | 527 | 551 | 1622
    PE | 296 | 286 | 278 | 860

OUTCOME MEASURES:

1. Primary Outcome: Adjudicated Composite of Symptomatic, Recurrent Venous Thromboembolism (VTE) or All-Cause Death During the Intended Treatment Period - Randomized Population With Imputation
Description: VTE included: nonfatal deep vein thrombosis (DVT) or nonfatal pulmonary embolism (PE). All index events, DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants with event) calculated as n/N (n=number of events; N=number of participants). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Composite endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. For missing endpoint data, participants were imputed as having had a primary efficacy outcome event.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with consent. Analyzed per randomized treatment assigned. (n) number of events=32, 34, 96 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively; number of events imputed=13, 20, 19, respectively. Confidence interval (CI) for event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0381 [0.0252 to 0.0510] | 0.0418 [0.0281 to 0.0556] | 0.1158 [0.0940 to 0.1376]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with VTE/all cause mortality to proportion of placebo participants with VTE/all cause mortality equal to 1.0. Participants with missing data were assumed to have experienced VTE/all cause mortality. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, Intent to treat (ITT) principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Hochberg adjusted p-value for superiority based on 2 hypotheses tests for apixaban 2.5mg group comparing with placebo group and for apixaban 5mg group comparing with placebo group; Risk Ratio (RR) = 0.3283, 95% CI 2-sided [0.2225 to 0.4844]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with VTE/all cause mortality to proportion of placebo participants with VTE/all cause mortality equal to 1.0. Participants with missing data were assumed to have experienced VTE/all cause mortality. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, Intent to treat principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.3615, 95% CI 2-sided [0.2475 to 0.5281]

2. Secondary Outcome: Adjudicated Composite of Recurrent, Symptomatic Venous Thromboembolism (VTE) or VTE-related Death During the Intended Treatment Period - Randomized Population With Imputation
Description: VTE includes nonfatal DVT or nonfatal PE. All index events, DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants with event) calculated as n/N (n=number of events; N=number of participants). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Composite endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. For missing endpoint data, participants were imputed as having had a primary efficacy outcome event.
Time Frame: Day 1 up to 12 Months
Population: ITT: all randomized participants with consent. Analyzed per randomized treatment assigned. (n) number of events=27, 34, 92 in apixaban 2.5 mg, 5 mg, placebo arms, respectively. Number of imputed events=13, 20, 19 in apixaban 2.5 mg, 5 mg, placebo arms, respectively. CI for single event rate was calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0321 [0.0202 to 0.0441] | 0.0418 [0.0281 to 0.0556] | 0.1110 [0.0896 to 0.1324]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with VTE/VTE-related death to proportion of placebo participants with VTE/ VTE-related death equal to 1.0. Participants with missing data were assumed to have experienced VTE/ VTE-related death. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.2891, 95% CI 2-sided [0.1902 to 0.4395]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.3774, 95% CI 2-sided [0.2577 to 0.5525]

3. Primary Outcome: Adjudicated Composite of Symptomatic, Recurrent Venous Thromboembolism (VTE) or All-Cause Death During the Intended Treatment Period - Randomized Population Without Imputation
Description: VTE included: nonfatal DVT or nonfatal PE. Event rate (proportion of participants with event) calculated as n/N (n=number of events; N=number of participants). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Composite endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for these endpoints; participants who had an event during the intended treatment period were counted. Confidence interval (CI) for single event rate was calculated based on the Wald asymptotic confidence limits.
Time Frame: Day 1 up to 12 months
Population: Intent to treat: all randomized participants with valid consent. Analyzed per randomized treatment assigned.(n)number of events = 19, 14, 77 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. All events were counted; no events were imputed.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0226 [0.0126 to 0.0327] | 0.0172 [0.0083 to 0.0262] | 0.0929 [0.0731 to 0.1126]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with VTE/all cause mortality to proportion of placebo participants with VTE/all cause mortality equal to 1.0. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, Intent to treat (ITT) principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.2422, 95% CI 2-sided [0.1476 to 0.3975]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.1861, 95% CI 2-sided [0.1062 to 0.3261]

4. Secondary Outcome: Adjudicated Composite of Recurrent, Symptomatic Venous Thromboembolism (VTE) or Cardio Vascular (CV) -Related Death During the Intended Treatment Period - Randomized Population With Imputation
Description: VTE includes nonfatal DVT or nonfatal PE. All index events, DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Composite endpoint included events that occurred any time from randomization until end of the intended treatment period, regardless of whether the participants were receiving drug treatment. Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. If there were missing endpoint data, participants were imputed as having had an efficacy outcome event.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with consent.(n)number of events=27, 34, 95 in apixaban 2.5 mg, 5 mg, placebo arms, respectively. The (n)number of imputed events were = 13, 20, 19 in apixaban 2.5 mg, 5 mg, placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
proportion of participants | 0.0321 [0.0202 to 0.0441] | 0.0418 [0.0281 to 0.0556] | 0.1146 [0.0929 to 0.1363]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with VTE/CV-related death to proportion of placebo participants with VTE/CV-related death equal to 1.0. Participants with missing data were assumed to have experienced VTE/CV-related death. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.2799, 95% CI 2-sided [0.1844 to 0.4247]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.3653, 95% CI 2-sided [0.2500 to 0.5338]

5. Secondary Outcome: Adjudicated Nonfatal Deep Vein Thrombosis (DVT) During the Intended Treatment Period - Randomized Population With Imputation
Description: DVT was adjudicated/confirmed by a central independent adjudication committee blinded to treatment and assessed by compression ultrasound and/or venography. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. Participants with missing endpoint information were classified as having had the efficacy event (imputation). Confidence interval (CI) for single event rate was calculated based on the Wald asymptotic confidence limits.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Analyzed per randomized treatment assigned. (n) number of events = 19, 28, 72 in apixaban 2.5 mg, 5 mg, placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0226 [0.0126 to 0.0327] | 0.0344 [0.0219 to 0.0470] | 0.0869 [0.0677 to 0.1060]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with nonfatal DVT to proportion of placebo participants with nonfatal DVT equal to 1.0. Participants with missing data were assumed to have experienced nonfatal DVT. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, Intent to treat (ITT) principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.2615, 95% CI 2-sided [0.1593 to 0.4292]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with nonfatal DVT to proportion of placebo participants with nonfatal DVT equal to 1.0. Participants with missing data were assumed to have experienced nonfatal DVT. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.3972, 95% CI 2-sided [0.2595 to 0.6079]

6. Secondary Outcome: Adjudicated Nonfatal Pulmonary Embolism (PE) During the Intended Treatment Period - Randomized Population With Imputation
Description: PE was adjudicated/confirmed by a central independent adjudication committee blinded to treatment and was assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. Participants with missing endpoint information were classified as having had the efficacy event (imputation). CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Analyzed per randomized treatment assigned. (n) number of events = 23, 25, 37 in apixaban 2.5 mg, 5 mg, placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0274 [0.0163 to 0.0384] | 0.0308 [0.0189 to 0.0426] | 0.0446 [0.0306 to 0.0587]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with nonfatal PE to proportion of placebo participants with nonfatal PE equal to 1.0. Participants with missing data were assumed to have experienced nonfatal PE. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p = 0.1084, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.6087, 95% CI 2-sided [0.3653 to 1.0145]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1329, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.6846, 95% CI 2-sided [0.4164 to 1.1257]

7. Secondary Outcome: Adjudicated Venous Thromboembolism (VTE) - Related Death During the Intended Treatment Period - Randomized Population With Imputation
Description: VTE-related death defined as: PE (based on objective diagnostic testing, autopsy), unexplained death (and VTE cannot be ruled out), sudden death (and VTE cannot be ruled out). DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. New/recurrent VTE, death, venous/arterial thromboembolic events, bleeding, thrombocytopenia, acute myocardial infarction and stroke were also adjudicated. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Participants with missing endpoint information were classified as having had the efficacy event (imputation).
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Analyzed per randomized treatment assigned. (n) number of events = 17, 24, 26 in apixaban 2.5 mg, 5 mg, placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0202 [0.0107 to 0.0298] | 0.0295 [0.0179 to 0.0412] | 0.0314 [0.0195 to 0.0432]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with VTE-related death to proportion of placebo participants with VTE-related death equal to 1.0. Participants with missing data were assumed to have experienced VTE-related death. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p = 0.3059, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.6470, 95% CI 2-sided [0.3543 to 1.1813]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.8288, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.9416, 95% CI 2-sided [0.5458 to 1.6245]

8. Secondary Outcome: Adjudicated Cardiovascular (CV)-Related Death During the Intended Treatment Period - Randomized Population With Imputation
Description: CV-related death was defined as myocardial infarction, stroke, or other specified cardiovascular event and were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. Participants with missing endpoint information were classified as having had the efficacy event (imputation). CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Analyzed per randomized treatment assigned. number of events (n)= 17, 24, 29 in the apixaban 2.5 mg, 5 mg, placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of Participants | 0.0202 [0.0107 to 0.0298] | 0.0295 [0.0179 to 0.0412] | 0.0350 [0.0225 to 0.0475]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with CV-related death to proportion of placebo participants with CV-related death equal to 1.0. Participants with missing data were assumed to have experienced CV-related death. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p = 0.1316, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.5794, 95% CI 2-sided [0.3215 to 1.0443]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.5288, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.8433, 95% CI 2-sided [0.4959 to 1.4341]

9. Secondary Outcome: Adjudicated All-Cause Death During the Intended Treatment Period - Randomized Population With Imputation
Description: DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. New/recurrent VTE, death, venous/arterial thromboembolic events, bleeding, thrombocytopenia, acute myocardial infarction and stroke were also adjudicated. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Participants with missing endpoint information were classified as having had the efficacy event (imputation). CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. (n) number of events = 22, 25, 33 in apixaban 2.5 mg, apixaban 5 mg, and placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0262 [0.0154 to 0.0370] | 0.0308 [0.0189 to 0.0426] | 0.0398 [0.0265 to 0.0531]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with all cause mortality to proportion of placebo participants with all cause mortality equal to 1.0. Participants with missing data were assumed to have experienced all cause mortality. Events occurring anytime during the intended treatment period (12 months) were included regardless of whether the participant was on treatment or not or whether the participant ever took drug, ie, ITT principle; Test type: Superiority or Other; p = 0.2361, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.6577, 95% CI 2-sided [0.3874 to 1.1169]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.3155, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.7708, 95% CI 2-sided [0.4631 to 1.2832]

10. Secondary Outcome: Number of Participants With an Adjudicated Symptomatic Nonfatal Venous Thromboembolism (VTE) Recurrence or Death (All Cause) During the Intended Treatment Period - Randomized Participants Without Imputation
Description: All index events, DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. First event category was the first primary event for each participant and each participant was counted once. CV-related death was presented excluding VTE-related death. In participants with event category, each participant was counted once in each event category but could have been counted in multiple categories. No imputation was done for these endpoints; participants who had an event during the intended treatment period were counted.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Analyzed per randomized treatment assigned. In first event (first primary event) each participant counted once. In event category, each participant was counted only once in each event category but could have been counted in multiple categories.
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
participants
  First event: Participants with nonfatal DVT | 6 | 7 | 53
  First event: Participants with nonfatal PE | 7 | 4 | 13
  First event: All-Cause Death | 6 | 3 | 11
  CV-related Death (included in all-cause total) | 0 | 0 | 3
  VTE-related Death (included in all-cause total) | 2 | 3 | 7
  Participants with event: nonfatal DVT | 6 | 8 | 53
  Participants with event: nonfatal PE | 8 | 4 | 15
  Participants with event: All cause death | 7 | 4 | 14

11. Secondary Outcome: Adjudicated Major Bleeding During the Treatment Period - Treated Population
Description: Major bleeding was adjudicated/confirmed by a central independent adjudication committee blinded to treatment and was defined as acute clinically overt bleeding: associated with a fall in hemoglobin of 2 grams per deciliter (g/dL) or more, or leading to a transfusion of 2 or more units of packed red blood cells or 1000 milliliters (mL) or more of whole blood, or in a critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal, or another critical organ; or is fatal. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Confidence interval (CI) for event rate was calculated based on the Wald asymptotic confidence limits. Treated population includes randomized participants who received at least one dose of study drug.
Time Frame: Day 1 up to 12 Months
Population: Treated population includes randomized participants who received at least one dose of study drug. (n) number of events = 2, 1, 4 in apixaban 2.5 mg, and 5 mg, and placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 811 | 826
Proportion of participants | 0.0024 [0.0000 to 0.0057] | 0.0012 [0.0000 to 0.0036] | 0.0048 [0.0001 to 0.0096]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with major bleeding to proportion of placebo participants with major bleeding equal to 1.0. Treated participants with at least one dose of study drug were included; Test type: Superiority or Other; p = 0.3925, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.4850, 95% CI 2-sided [0.0891 to 2.6391]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with major bleeding to proportion of placebo participants with major bleeding equal to 1.0. Participants treated with at least one dose of study drug were included; Test type: Superiority or Other; p = 0.3551, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.2457, 95% CI 2-sided [0.0269 to 2.2437]

12. Secondary Outcome: Adjudicated Composite of Major/Clinically Relevant Non-major Bleeding During the Treatment Period - Treated Participants
Description: Major bleeding and clinically relevant non-major bleeding were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. Major bleeding was defined as acute clinically overt bleeding: associated with a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of 2 or more units of packed red blood cells or 1000 mL or more of whole blood, or in a critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal, or another critical organ or is fatal. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). CI for single event rate was calculated based on the Wald asymptotic confidence limits. Treated population includes randomized participants who received at least one dose of study drug.
Time Frame: Day 1 up to 12 Months
Population: Treated participants were those who received at least 1 dose of study drug. (n)number of events = 27, 35, 22 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 811 | 826
proportion of participants | 0.0321 [0.0202 to 0.0441] | 0.0432 [0.0292 to 0.0571] | 0.0266 [0.0157 to 0.0376]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg; Null hypothesis is relative risk proportion of apixaban participants with major/clinically relevant non-major bleeding to proportion of placebo participants with major/clinically relevant non-major bleeding equal to 1.0; Test type: Superiority or Other; p = 0.5148, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.2027, 95% CI 2-sided [0.6897 to 2.0975]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.1412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.6160, 95% CI 2-sided [0.9554 to 2.7336]

13. Secondary Outcome: Adjudicated Clinically Relevant Non-major Bleeding During the Treatment Period - Treated Participants
Description: Non-major clinically relevant bleeding was adjudicated/confirmed by a central independent adjudication committee blinded to treatment and defined as: acute clinically overt bleeding compromising hemodynamics; leading to hospitalization; traumatic subcutaneous hematoma; intramuscular hematoma; epistaxis that lasted for more than 5 minutes, was repetitive or led to an intervention; spontaneous gingival bleeding (or lasting more than 5 minutes); spontaneous hematuria (macroscopic or lasted more than 24 hours after instrumentation of the urogenital tract); macroscopic gastrointestinal hemorrhage (including at least 1 episode of melena or hematemesis (if clinically apparent with positive results on a fecal occult-blood test); rectal blood loss. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Time Frame: Day 1 up to 12 months
Population: Treated population includes randomized participants who received at least one dose of study drug. (n)number of events = 25, 34, 19 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 811 | 826
Proportion of participants | 0.0298 [0.0183 to 0.0413] | 0.0419 [0.0281 to 0.0557] | 0.0230 [0.0128 to 0.0332]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with clinically relevant non-major bleeding to proportion of placebo participants with clinically relevant non-major bleeding equal to 1.0; Test type: Superiority or Other; p = 0.3932, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.2928, 95% CI 2-sided [0.7158 to 2.3348]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0621, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.8235, 95% CI [1.0470 to 3.1760]

14. Secondary Outcome: Adjudicated Clinically Relevant Minor Bleeding During the Treatment Period - Treated Participants
Description: All bleeding events were reviewed by the central independent adjudication committee blinded to treatment and classified as major bleeding, clinically relevant non-major bleeding, minor bleeding or no bleeding. If event was not major or clinically relevant non-major, it was judged to be minor. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Confidence interval (CI) for single event rate was calculated based on the Wald asymptotic confidence limits. Treated population includes randomized participants who received at least one dose of study drug.
Time Frame: Day 1 up to 12 months
Population: Treated population includes randomized participants who received at least one dose of study drug. (n)number of events = 75, 98, 58 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 811 | 826
Proportion of participants | 0.0893 [0.0700 to 0.1086] | 0.1208 [0.0984 to 0.1433] | 0.0702 [0.0528 to 0.0876]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with minor bleeding to proportion of placebo participants with minor bleeding equal to 1.0; Test type: Superiority or Other; p = 0.1691, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.2579, 95% CI 2-sided [0.9064 to 1.7457]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.6971, 95% CI 2-sided [1.2468 to 2.3102]

15. Secondary Outcome: Adjudicated Total Bleeding During the Treatment Period - Treated Participants
Description: All bleeding events were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. Total bleeding was defined as any major, clinically relevant non-major, or minor bleeding. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). CI for single event rate was calculated based on the Wald asymptotic confidence limits. Treated population includes randomized participants who received at least one dose of study drug.
Time Frame: Day 1 up to 12 months
Population: Treated population includes randomized participants who received at least one dose of study drug. (n) number of events = 94, 121, 74 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 811 | 826
Proportion of participants | 0.1119 [0.0906 to 0.1332] | 0.1492 [0.1247 to 0.1737] | 0.0896 [0.0701 to 0.1091]
Statistical Analysis 1: Comparison: Apixaban 2.5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with total bleeding to proportion of placebo participants with total bleeding equal to 1.0. Total bleeding was defined as any major, clinically relevant non-major, or minor bleeding; Test type: Superiority or Other; p = 0.1466, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.2374, 95% CI 2-sided [0.9276 to 1.6507]
Statistical Analysis 2: Comparison: Apixaban 5 mg vs Placebo; Null hypothesis is relative risk proportion of apixaban participants with total bleeding to proportion of placebo participants with total bleeding equal to 1.0. Total bleeding is any major, clinically relevant non-major, or minor bleeding; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.6468, 95% CI 2-sided [1.2552 to 2.1606]

16. Secondary Outcome: Adjudicated Composite of Recurrent, Symptomatic Venous Thromboembolism (VTE) or Venous Thromboembolism-related Death During the Intended Treatment Period - Randomized Population Without Imputation
Description: VTE related death defined as PE (based on objective diagnostic testing, autopsy), unexplained death (and VTE cannot be ruled out), sudden death (and VTE cannot be ruled out). DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. New/recurrent VTE and death, were also adjudicated. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for these endpoints.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 14, 14, 73 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
proportion of participants | 0.0167 [0.0080 to 0.0253] | 0.0172 [0.0083 to 0.0262] | 0.0881 [0.0688 to 0.1073]

17. Secondary Outcome: Adjudicated Composite of Recurrent, Symptomatic Venous Thromboembolism (VTE) or Cardio Vascular (CV) - Related Death During the Intended Treatment Period - Randomized Population Without Imputation
Description: CV-related death was defined as myocardial infarction, stroke, or other specified cardiovascular event. Index events of DVT and/or PE, along with myocardial infarction and stroke were adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Composite endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for these endpoints; participants who had an event during the intended treatment period were counted.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 14, 14, 76 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
proportion of participants | 0.0167 [0.0080 to 0.0253] | 0.0172 [0.0083 to 0.0262] | 0.0917 [0.0720 to 0.1113]

18. Secondary Outcome: Adjudicated Nonfatal Deep Vein Thrombosis (DVT) During the Intended Treatment Period - Randomized Population Without Imputation
Description: DVT was adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for this endpoint; participants who had an event during the intended treatment period were counted.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 6, 8, 53 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
proportion of participants | 0.0071 [0.0014 to 0.0128] | 0.0098 [0.0031 to 0.0166] | 0.0639 [0.0473 to 0.0806]

19. Secondary Outcome: Adjudicated Nonfatal Pulmonary Embolism (PE) During the Intended Treatment Period - Randomized Population Without Imputation
Description: PE was adjudicated/confirmed by a central independent adjudication committee blinded to treatment: PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for this endpoint; participants who had an event during the intended treatment period were counted.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 8, 4, 15 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0095 [0.0030 to 0.0161] | 0.0049 [0.0001 to 0.0097] | 0.0181 [0.0090 to 0.0272]

20. Secondary Outcome: Adjudicated Venous Thromboembolism (VTE)- Related Death During the Intended Treatment Period - Randomized Population Without Imputation
Description: VTE related death defined as PE (based on objective diagnostic testing, autopsy), unexplained death (and VTE cannot be ruled out), sudden death (and VTE cannot be ruled out). DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. New/recurrent VTE, and death, were also adjudicated. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for this endpoint.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 2, 3, 7 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0024 [0.0000 to 0.0057] | 0.0037 [0.0000 to 0.0079] | 0.0084 [0.0022 to 0.0147]

21. Secondary Outcome: Adjudicated Cardio Vascular (CV)-Related Death During the Intended Treatment Period - Randomized Population Without Imputation
Description: CV-related death was defined as myocardial infarction, stroke, or other specified cardiovascular event and these were adjudicated/confirmed by a central independent adjudication committee blinded to treatment. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for this endpoint; participants who had an event during the intended treatment period were counted.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 2, 3, 10 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0024 [0.0000 to 0.0057] | 0.0037 [0.0000 to 0.0079] | 0.0121 [0.0046 to 0.0195]

22. Secondary Outcome: Adjudicated All-Cause Death During the Intended Treatment Period - Randomized Population Without Imputation
Description: DVT and/or PE were adjudicated/confirmed by a central independent adjudication committee blinded to treatment: DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. New/recurrent VTE, death, venous/arterial thromboembolic events, bleeding, thrombocytopenia, acute myocardial infarction and stroke were also adjudicated. Event rate is proportion of participants with event; calculated as n/N (n=number of events; N=number of participants). Intended treatment period was defined as the longer of the dosing period plus 2 days or 355 days. Endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received. No imputation was done for this endpoint; participants who had an event during the intended treatment period were counted.
Time Frame: Day 1 up to 12 Months
Population: Intent to treat: all randomized participants with valid consent. Participants analyzed per randomized treatment assigned. (n) number of events = 7, 4, 14 in apixaban 2.5 mg, 5 mg, and placebo arms, respectively. CI for single event rate was calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg | Placebo
Number analyzed (Participants) | 840 | 813 | 829
Proportion of participants | 0.0083 [0.0022 to 0.0145] | 0.0049 [0.0001 to 0.0097] | 0.0169 [0.0081 to 0.0257]

ADVERSE EVENTS:
Time Frame: Day 1 up to 12 months
Groups:
- Apixaban 2.5mg: Participants received 2.5 mg oral tablet apixaban BID
- Apixaban 5mg: Participants received 5 mg oral tablet apixaban BID
- Placebo: Participants received oral tablet of placebo BID
Arm/Group | Apixaban 2.5mg | Apixaban 5mg | Placebo
Serious Adverse Events (participants affected / at risk) | 112/840 | 107/811 | 158/826
Other Adverse Events (participants affected / at risk) | 341/840 | 305/811 | 318/826
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 2.5mg (N=840) | Apixaban 5mg (N=811) | Placebo (N=826)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 3 | 2
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 3 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 1 | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1 | 4
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 0 | 1
EXTRASYSTOLES (Cardiac disorders) | 1 | 0 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 3 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 3
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 1 | 0
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 1 | 0 | 0
OTOSCLEROSIS (Ear and labyrinth disorders) | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 2
THYROIDITIS (Endocrine disorders) | 0 | 0 | 1
CATARACT (Eye disorders) | 1 | 0 | 0
EYE HAEMORRHAGE (Eye disorders) | 0 | 0 | 2
MACULAR OEDEMA (Eye disorders) | 1 | 0 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 1 | 0 | 0
RETINAL VEIN OCCLUSION (Eye disorders) | 1 | 0 | 0
RETINAL VEIN THROMBOSIS (Eye disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 0 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 2 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1 | 0
ILEUS (Gastrointestinal disorders) | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0
POLYP COLORECTAL (Gastrointestinal disorders) | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1
DEATH (General disorders) | 0 | 0 | 2
FATIGUE (General disorders) | 0 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 1 | 0
SUDDEN DEATH (General disorders) | 0 | 1 | 3
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 1
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 2 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 3 | 0 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 | 2 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 1
AMYLOIDOSIS (Immune system disorders) | 1 | 0 | 0
ANTIPHOSPHOLIPID SYNDROME (Immune system disorders) | 0 | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 2 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 2 | 0 | 2
DIVERTICULITIS (Infections and infestations) | 1 | 1 | 0
EMPYEMA (Infections and infestations) | 0 | 1 | 0
ENCEPHALITIS MENINGOCOCCAL (Infections and infestations) | 0 | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 0 | 0
HAEMATOMA INFECTION (Infections and infestations) | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 2
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
ORCHITIS (Infections and infestations) | 0 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 1
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 5 | 3 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 2 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 3 | 1
SALPINGITIS (Infections and infestations) | 1 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 2 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1
TONSILLITIS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1
VIRAL SINUSITIS (Infections and infestations) | 1 | 0 | 0
ACCIDENTAL EXPOSURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 | 1 | 0
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
HEAT EXHAUSTION (Injury, poisoning and procedural complications) | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1 | 0
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 1
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
BIOPSY BONE (Investigations) | 0 | 0 | 1
COAGULATION TIME PROLONGED (Investigations) | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
JOINT ANKYLOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
LIGAMENT DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
BENIGN PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
CARCINOID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
METASTATIC BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
NON-HODGKIN'S LYMPHOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
RECTAL CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
VOCAL CORD NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1 | 3
CONVULSION (Nervous system disorders) | 1 | 1 | 0
DEMYELINATING POLYNEUROPATHY (Nervous system disorders) | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 0 | 1
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 | 0 | 0
FEBRILE CONVULSION (Nervous system disorders) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 2 | 0
HEMIANOPIA HOMONYMOUS (Nervous system disorders) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 1 | 2
MIGRAINE (Nervous system disorders) | 1 | 0 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 | 0 | 1
OPTIC NEURITIS (Nervous system disorders) | 0 | 1 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 2 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 2
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 1
ALCOHOLISM (Psychiatric disorders) | 1 | 0 | 0
DELIRIUM (Psychiatric disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1
DRUG DEPENDENCE (Psychiatric disorders) | 0 | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 2 | 2
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1 | 3
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0
URETERIC STENOSIS (Renal and urinary disorders) | 0 | 0 | 2
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
ALLERGIC GRANULOMATOUS ANGIITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 20
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
MISCARRIAGE OF PARTNER (Social circumstances) | 0 | 0 | 1
PREGNANCY OF PARTNER (Social circumstances) | 0 | 1 | 1
ABORTION INDUCED (Surgical and medical procedures) | 0 | 0 | 1
HOSPITALISATION (Surgical and medical procedures) | 0 | 2 | 1
ANEURYSM (Vascular disorders) | 0 | 0 | 1
ARTERIAL DISORDER (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 9 | 40
EMBOLISM VENOUS (Vascular disorders) | 0 | 0 | 1
FEMORAL ARTERY EMBOLISM (Vascular disorders) | 1 | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 1
MALIGNANT HYPERTENSION (Vascular disorders) | 1 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 1 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 1
THROMBOSIS (Vascular disorders) | 1 | 0 | 0
VARICOPHLEBITIS (Vascular disorders) | 0 | 1 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 3
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 2.5mg (N=840) | Apixaban 5mg (N=811) | Placebo (N=826)
CONSTIPATION (Gastrointestinal disorders) | 18 | 12 | 14
DIARRHOEA (Gastrointestinal disorders) | 37 | 24 | 24
NAUSEA (Gastrointestinal disorders) | 20 | 18 | 20
FATIGUE (General disorders) | 17 | 14 | 10
OEDEMA PERIPHERAL (General disorders) | 28 | 25 | 33
BRONCHITIS (Infections and infestations) | 24 | 30 | 13
INFLUENZA (Infections and infestations) | 18 | 20 | 20
NASOPHARYNGITIS (Infections and infestations) | 41 | 31 | 40
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 18 | 18
URINARY TRACT INFECTION (Infections and infestations) | 28 | 30 | 34
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 26 | 20 | 21
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 32 | 21 | 22
BACK PAIN (Musculoskeletal and connective tissue disorders) | 27 | 45 | 24
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 21 | 16 | 13
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 44 | 52 | 54
DIZZINESS (Nervous system disorders) | 20 | 18 | 15
HEADACHE (Nervous system disorders) | 44 | 41 | 42
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 21 | 18
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18 | 15 | 19
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 13 | 27 | 8
RASH (Skin and subcutaneous tissue disorders) | 18 | 8 | 12
DEEP VEIN THROMBOSIS (Vascular disorders) | 12 | 8 | 23
HYPERTENSION (Vascular disorders) | 34 | 19 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.